CLINICAL TRIAL: NCT03066648
Title: Phase 1b, Multi-arm, Open-label Study of PDR001 and/or MBG453 in Combination With Decitabine in Patients With Acute Myeloid Leukemia or High Risk Myelodysplastic Syndrome
Brief Title: Study of PDR001 and/or MBG453 in Combination With Decitabine in Patients With AML or High Risk MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001X2105; 2016-005060-33 (EudraCT Number)
Record Dates: First submitted 2017-02-18; First posted 2017-02-28 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Preleukemia; Bone Marrow Diseases; Hematologic Diseases; Chronic Myelomonocytic Leukemia
Keywords: Acute Myeloid Leukemia; Myelodysplastic syndromes; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Preleukemia; Bone Marrow Diseases; Hematologic Diseases; Leukemia, Myelomonocytic, Chronic | interventions — Decitabine; spartalizumab; sabatolimab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Decitabine and PDR001 (Experimental): Decitabine in combination with PDR001
  Interventions: Drug: Decitabine; Drug: PDR001
- Decitabine and MBG453 (Experimental): Decitabine in combination with MBG453
  Interventions: Drug: Decitabine; Drug: MBG453
- Decitabine, PDR001 and MBG453 (Experimental): Decitabine in combination with PDR001 and MBG453
  Interventions: Drug: Decitabine; Drug: PDR001; Drug: MBG453
- MBG453 (Experimental): MBG453 alone
  Interventions: Drug: MBG453
- MBG453 and PDR001 (Experimental): MBG453 in combination with PDR001
  Interventions: Drug: PDR001; Drug: MBG453
- Azacitidine and MBG453 (Experimental): Azacitidine in combination with MBG453
  Interventions: Drug: MBG453; Drug: Azacitidine

INTERVENTIONS:
Drug: Decitabine — Decitabine is a cytidine deoxynucleoside analogue that selectively inhibits DNA methyltransferases at low doses, resulting in gene promoter hypomethylation.
  Other Names: 5-aza-2'-deoxycytidine
  Arms: Decitabine and MBG453; Decitabine and PDR001; Decitabine, PDR001 and MBG453
Drug: PDR001 — PDR001 is a high-affinity, ligand-blocking, humanized IgG4 monoclonal antibody directed against PD-1 that blocks the binding of PD-L1 and PD-L2.
  Other Names: spartalizumab
  Arms: Decitabine and PDR001; Decitabine, PDR001 and MBG453; MBG453 and PDR001
Drug: MBG453 — MBG453 is a high-affinity, humanized anti-TIM-3 IgG4 monoclonal antibody which blocks the binding of TIM-3 to phosphatidylserine (PtdSer).
  Other Names: sabatolimab
  Arms: Azacitidine and MBG453; Decitabine and MBG453; Decitabine, PDR001 and MBG453; MBG453; MBG453 and PDR001
Drug: Azacitidine — Azacitidine (5-azacytidine) is a cytidine nucleoside analogue that selectively inhibits DNA methyltransferases at low doses, resulting in gene promoter hypomethylation
  Other Names: 5-azacytidine
  Arms: Azacitidine and MBG453

SUMMARY:
To characterize the safety and tolerability of 1) MBG453 as a single agent or in combination with PDR001 or 2) PDR001 and/or MBG453 in combination with decitabine or azacitidine in AML and intermediate or high- risk MDS patients, and to identify recommended doses for future studies.

DETAILED DESCRIPTION:
This is a phase 1b, multi-arm, open-label study in patients with acute myeloid leukemia (AML) or intermediate or high risk myelodysplastic syndrome (MDS). Patients with myelodysplastic-myeloproliferative neoplasms (MDS/MPN), including chronic myelomonocytic leukemia (CMML) could also be enrolled.

The study was comprised of six arms as described below. Arms 1-3 enrolled patients with newly diagnosed AML who were planned for non-intensive chemotherapy, relapsed/refractory (R/R) AML, or intermediate or high-risk MDS.

* Arm 1: Evaluation of a fixed dose of the standard of care agent decitabine in combination with fixed dose PDR001.
* Arm 2: Evaluation of a fixed dose of the standard of care agent decitabine in combination with escalating dose MBG453.
* Arm 3: Evaluation of a fixed dose of the standard of care agent decitabine in combination with fixed dose PDR001 and escalating dose MBG453.

Arms 4-5 enrolled patients with R/R AML or intermediate or high-risk MDS who had failed hypomethylating agent therapy.

* Arm 4: Evaluation of an escalating dose of MBG453
* Arm 5: Evaluation of an escalating dose of MBG453 in combination with fixed dose PDR001 Arm 6 enrolled patients with newly diagnosed AML who were planned for non-intensive chemotherapy, or intermediate or high-risk MDS.
* Arm 6: Evaluation of a fixed dose of the standard of care agent azacitidine in combination with an escalating dose of MBG453.

Patients received the assigned treatment until disease progression, unacceptable toxicity, start of a new anti-neoplastic therapy, discontinuation at the discretion of the investigator or patient, lost to follow-up, death, or the study termination, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures
2. Male or female patients ≥ 18 years of age who present with one of the following:

   Arms 1-3:
   * Relapsed/refractory AML following ≥1 prior therapies who have relapsed or exhibited refractory disease (primary failure) and are deemed by the investigator not to be candidates for standard therapy, including re-induction with cytarabine or other established chemotherapy regimens for patients with AML (patients who are suitable for standard re-induction chemotherapy or hematopoietic stem cell transplantation and willing to receive it are excluded)
   * Newly diagnosed AML patients who are suitable for treatment with decitabine (patients who are suitable for standard induction chemotherapy or hematopoietic stem cell transplantation and willing to receive it are excluded)
   * Intermediate or high risk MDS or MDS/MPN including CMML (patients who are suitable for standard re-induction chemotherapy or hematopoietic stem cell transplantation and willing to receive it are excluded)

   Arms 4-5:
   * Refractory / relapsed AML following ≥1 prior therapies (Arms 4a & 5a)
   * Intermediate or high risk MDS or MDS/MPN including CMML who have failed hypomethylating agent therapy (Arms 4b & 5b) (Note: hypomethylating agent failure is defined as progressive disease on hypomethylating agent therapy or lack of clinically meaningful response as deemed by investigator after at least 4 cycles of hypomethylating agent therapy.)

   Arm 6:
   * Newly diagnosed AML patients who are suitable for treatment with azacitidine (patients who are suitable for standard induction chemotherapy or hematopoietic stem cell transplantation and willing to receive it are excluded) (Arm 6a)
   * Intermediate or high-risk MDS or MDS/MPN including CMML (patients who are suitable for standard induction chemotherapy or hematopoietic stem cell transplantation and willing to receive it are excluded) (Arm 6b)
3. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
4. Patient must be a candidate for serial bone marrow aspirate and/or biopsy according to the institutions guidelines and be willing to undergo a bone marrow aspirate and/biopsy at screening, during and at the end of therapy on this study. Exceptions may be considered after documented discussion with Novartis.
5. Arms 1-3: Patients must be fit for standard treatment with decitabine as determined by the investigator and as per local decitabine package insert.
6. Arm 6: Patients must be fit for standard treatment with azacitidine as determined by the investigator and as per the local azacitidine package insert.

Exclusion Criteria:

1. Arms 1-3 or Arm 6: Patients who have received prior hypomethylating agent treatment for AML or MDS.
2. Patients with active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur should not be excluded.
3. History of, or current drug-induced interstitial lung disease or pneumonitis grade ≥ 2.
4. Patients who discontinued prior PD-1 or PD-L1 directed therapy due to a treatment related toxicity should not be included in the PDR001 containing arms of the study. Patients previously exposed to anti-PD-1/PD-L1 treatment who are adequately treated for skin rash or with replacement therapy for endocrinopathies should not be excluded.
5. Systemic antineoplastic therapy (including cytotoxic chemotherapy, alphainterferon, kinase inhibitors or other targeted small molecules, and toxinimmunoconjugates) or any experimental therapy within 14 days or 5 half-lives, whichever is shorter, before the first dose of study treatment.
6. Systemic chronic corticosteroid therapy (>10 mg/day prednisone or equivalent) or any immunosuppressive therapy within 7 days of first dose of study treatment. Topical, inhaled, nasal and ophthalmic steroids are allowed.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Safety of MBG453 single agent treatment or MBG453 in combination with PDR001 or PDR001 and/or MBG453 in combination with decitabine or azacitidine. | 24 months
  Incidence and severity of AEs and SAEs
Incidence of Dose Limiting Toxicities (DLTs) | 2 months
  The incidence of DLTs during the first two cycles of treatment with MBG453 in combination with PDR001 or PDR001 and/or MBG453 in combination with decitabine.
Incidence of Dose Limiting Toxicities (DLTs) | 1 month
  The incidence of DLTs during the first cycle of MBG453 single agent treatment or during the first two cycles of treatment with MBG453 in combination with PDR001 or PDR001 and/or MBG453 in combination with decitabine.
Tolerability of MBG453 single agent treatment or MBG453 in combination with PDR001 or PDR001 and/or MBG453 in combination with decitabine or azacitidine. | 24 months
  Incidence and severity of AEs and SAEs

SECONDARY OUTCOMES:
AUC of PDR001, MBG453, decitabine and azacitidine. | 24 months
  AUC
Cmax of PDR001, MBG453, decitabine and azacitidine | 24 months
  Cmax
Tmax of PDR001, MBG453, decitabine and azacitidine | 24 months
  Tmax
Half-life of PDR001, MBG453, decitabine and azacitidine | 24 months
  Half-life
Overall Response Rate (ORR) | 24 months
  Determine ORR in each arm of the study
Best Overall Response (BOR) | 24 months
  Determine BOR in each arm of the study
Progression Free Survival (PFS) | 24 months
  Determine PFS in each arm of the study
Time to Progression (TTP) | 24 months
  Determine TTP in each arm of the study
Duration of Response (DOR) | 24 months
  Determine DOR in each arm of the study
Number of participants with anti-PDR001 and anti-MBG453 antibodies | 24 months
  Presence of anti-PDR001 and anti-MBG453 antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Oregon Health Sciences University Main Center, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Helsinki, Finland
- Novartis Investigative Site, Marseille, France
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Jena
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18210
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2288